CLINICAL TRIAL: NCT01870115
Title: Phase 1 Study of Combination Strontium, Melatonin and Nutritional Co-factors on Bone Health and Quality of Life in Postmenopausal Women With Osteopenia
Brief Title: Melatonin-Micronutrients for Osteopenia Treatment Study
Acronym: MOTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duquesne University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Grant Protocol Number 13-59
Record Dates: First submitted 2013-06-03; First posted 2013-06-05 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2017-02

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Melatonin; Strontium Citrate; Osteoporosis; Osteopenia
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Dietary Fiber; Melatonin

STUDY DESIGN:
Intervention Model Description: Melatonin (5mg), strontium (citrate; 450mg) vitamin D3 (2000IU)and vitamin K2 (MK7; 60mcg)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber pill (Placebo Comparator): 2 plant fiber pills taken p.o. (by mouth) nightly for one year
  Interventions: Dietary Supplement: Fiber Pill
- strontium/melatonin/Vitamins K2 and D3 (Active Comparator): 2 pills taken p.o. (by mouth) nightly for one year. Each pill contains strontium citrate (225 mg), melatonin (2.5 mg), Vitamin K2 (MK7) (30 mcg) and Vitamin D3 (1000 IU)
  Interventions: Dietary Supplement: Melatonin, Strontium citrate, Vitamins D3 and K2

INTERVENTIONS:
Dietary Supplement: Fiber Pill — This fiber pill has been manufactured to mimic the pill that contains the dietary supplements melatonin (M), strontium citrate (S), vitamin D3 (D) and vitamin K2 (K) in appearance but does not contain the supplements
  Arms: Fiber pill
Dietary Supplement: Melatonin, Strontium citrate, Vitamins D3 and K2 — Each pill has been manufactured to contain the dietary supplements 2.5mg melatonin (M), 225mg strontium citrate (S), 1000IU vitamin D3 (D) and 30mcg vitamin K2 (K)
  Arms: strontium/melatonin/Vitamins K2 and D3

SUMMARY:
The investigators' long-term goal is to employ novel methods to improve bone formation and bone density in women (and men) with osteopenia or osteoporosis while also decreasing signs and symptoms of degenerative joint and disc disease that commonly accompany bone loss as well as improve quality of life (QOL). These conditions generally begin silently as early as the menopause transition and progress to osteopenia and osteoporosis during the post-menopausal years in aging women. The investigators also envision this will be beneficial in aging andropausal men with these conditions. The investigators postulate that melatonin in novel combination with other natural bone-protective agents may act in a "chronosynergy" manner to prevent and correct these perturbations, reducing the risk of bone fractures, and lessening the stiffness and pain associated with bone, joint and cartilage degeneration and improving quality of life (QOL). The objective here, which is the investigators' next step in pursuit of our goal, is to assess the efficacy of an alternative therapy that uses a novel combination of bone-forming agents, melatonin, strontium (citrate)/ vitamin K2 (MK7), and vitamin D3 on bone health in a postmenopausal population. Melatonin is a novel alternative to current treatment(s) because it has multiple bone-protective and sleep-promoting activities within the body, and it is relatively safe so it can be used in an aging population without untoward side effects; strontium and vitamin D3 are shown to enhance bone mineralization and improve post-menopausal osteoporosis. The project goal is to identify if this combination therapy improves bone health and QOL compared to women taking placebo. The investigators' central hypothesis is that combination therapy using melatonin, strontium, vitamin K2, and vitamin D3 will improve bone health and overall QOL in postmenopausal women not taking this regimen by reducing osteoclast activity and increasing osteoblast activity and by improving subjective measures of stress, anxiety, depression and menopause-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal
* must be osteopenic (T-score between -2.5 and -1)
* willingness to participate in the 12-month study
* willingness to undergo testing of bone turnover markers before and after the drug therapies
* willingness to provide a self-assessment on quality of life throughout the program
* willingness to take their treatments right before bed
* willingness to not to consume alcohol with this medication

Exclusion Criteria:

* women in whom osteopenia is a result of some other known process (e.g. hyperparathyroidism, metastatic bone disease, multiple myeloma or chronic steroid use).
* women on osteoporotic drugs, hypnotics, CYP1A2 inhibiting drugs, fluvoxamine
* women with severe sleep apnea, severe COPD and those with moderate or severe hepatic or renal impairment.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-08; Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
Changes in bone mineral density from baseline to one year following treatment | One year

CONTACTS AND LOCATIONS:
Overall Officials: Paula A Witt-Enderby, PhD, Principal Investigator — Duquesne University; Mark Swanson, ND, Principal Investigator — Private Practice
Locations (1):
- Duquesne University Center for Pharmacy Care, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Publication — http://www.aging-us.com/article/101158